CLINICAL TRIAL: NCT04835090
Title: Comparison of the State Transition, Psychometric Attributes and Feasibility of Three Frailty Screening Tools in Community-dwelling Elderly
Brief Title: Comparison of Three Frailty Screening Tools
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Wei Gong Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hung-Ru Lin, PhD, RN, Professor, School of Nursing & Dean of Academic Affairs, National Taipei University of Nursing and Health Sciences
Other Study IDs: 200836
Record Dates: First submitted 2021-02-22; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Frailty
Keywords: frailty; transition; psychometric attributes; feasibility; screening; community-dwelling; elderly
MeSH Terms: conditions — Frailty | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: screening test — using three screening tools

SUMMARY:
The financial health care and social impact of the frailty of the elderly is an important issue for preventive health care in various countries around the world. The Taiwan government launched the long-term care 10-year plan version 2.0 in 2017 and expanded service target with older people with frailty as a service need. There is no consensus on the definition of frailty. However, there are many existing frailty screening instruments. It is very important to choose accurate and simple and rapid tools for screening to reduce the extra medical costs caused by negative outcomes of frailty. The primary purpose of this study is to understand the transition changes of the elderly in the community during the six months of frail state (robust, pre-frail, frail), and examine the validity of the frailty, physical function (handgrip strength, walking speed) to predict negative outcomes (falls, institutionalization/hospitalization), and will be compared with the results of three frailty screening tools. The secondary purpose is to compare the feasibility (screening time, screening completion rate, equipment and space) of the three tools for the frailty screening of the elderly in the community.

DETAILED DESCRIPTION:
This is a prospective study with six month follow-up among community-dwelling elderly aged 65 or older. Agreement between instruments, Frail state transition changes, feasibility, internal consistency, concurrent and predictive validity, convergent validity of instruments will be evaluated and compared. The participants' recruitment strategies will be through referrals by the personnel in outpatient department in a hospital, community care centers, health centers, C tiers of community care service system, love angel stations etc. We focused on three available instruments based on literature review and expert opinions for community-dwelling elderly care: Kihon Checklist (KCL), Study of Osteoporotic Fractures (SOF), and frailty phenotype (FP) screening tools. Using G-power3.1 for sample size estimation, 80 subjects will be needed. Based on the estimated loss rate is 30%, so 110 participants need to be recruited.

The screening sequence of this research will carry out with the Randomization block. There are six sequence combinations with three frailty screening tools. The researcher read the questionnaire one by one item, and then will fill the participants' answers into the data collection sheets. The physical function test is performed by the researcher.

This study was approved by the institutional Review Board. All participants will be asked to complete written informed consent. The statistical method adopts multivariate repeated measure analysis to detect the transition of frailty state. The area under the curve (AUC) will be used to examine the predictive ability on body function (grip strength, walking speed) and negative outcomes (falls, hospitalization) of the three frailty screening tools.

The anticipated benefits of this study will include (1) clinical practice: provide the screening time, completion rate, reliability and validity of the frailty screening tools to clinical health care professionals with reference to the selection of frailty screening tools for the community-dwelling elderly. Predicting the cut-off point of screening for falls or institutionalization/hospitalization of elderly people in the community can be used in nursing clinical practice to explain the screening results and risk assessment of falls and hospitalization to patients to prevent or delay the frailty progress. (2) academic research: provide a six-month observation of the changes in the frailty status of the elderly in the community in Taiwan, increase the understanding of the frailty transition of the elderly in the community, and identify frailty screening tools that have better prediction of physical functions and negative results. (3) National development: The results of this study are provided to the government as a reference for optimizing Taiwan's long-term care 2.0 policy formulation.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 65 years and older with community-dwelling in Taoyuan and Hsinchu city, Miaoli county
2. Communicate with Mandarin, Taiwanese, or Hakka
3. Agreement to participant the frailty screening three times within half a year after explanation, and have signed an informed consent.

Exclusion Criteria:

1. Living in a hospital or nursing home.
2. Dementia.
3. Bedridden or terminal illness.
4. Taking drugs for Alzheimer's disease or antidepressant drugs.
5. Stroke or upper or lower limb surgery in the past three months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-dwelling elderly aged 65 or older referral by the personnel in outpatient department in a hospital, community care centers, activity centers, health centers, C tiers of community care service system, health stations, love angel stations, long-term care centers, and community development associations.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Change in Frailty Phenotype (FP) | This will be measured at baseline, three months and six months.
  The FP measurement tool consists five items (yes/no) which includes handgrip strength measured via a dynamometer (in kilograms), self-reported weight loss, self-reported exhaustion, 5 meter usual gait speed (in seconds), and physical activity level measured by the Taiwan International Physical Activity Questionnaire Short Form (Taiwanese version of the IPAQ), which was used to calculate calorie consumption. The number of criteria (a 6-level ordinal variable ranging from 0 to 5) is categorized into a 3-level variable depicting robust (none of the criteria), pre-frail (one or two criteria) and frail (three or more criteria).
Change in Study of Osteoporotic Fractures (SOF) | This will be measured at baseline, three months and six months.
  The SOF consists three items (yes/no) which includes weight loss (unintentional); inability to rise from a chair 5 times without the use of arms; and reduced energy level. Frail status was defined as robust (none of components), prefrail (one component), and frail (two or more components).
Change in Kihon Checklist (KCL) | This will be measured at baseline, three months and six months.
  The KCL consists of 25 items (yes/no) divided into seven domains: physical strength, nutrition, eating, socialization, memory, mood; each domain is rated on a pass (0)/fail (1) basis, and the sum of all indices ranges from 0 (no frailty) to 25 (severe frailty); a higher score indicates worse functioning. Frailty status was defined as robust (0-3 scores), prefrail (4-7 scores), and frail (8 scores or more ).
Change in Handgrip Strength | This will be measured at baseline, three months and six months.
  handgrip strength measured via a dynamometer (in kilograms)
Change in Gait Speed | This will be measured at baseline, three months and six months.
  5 meter usual gait speed (in seconds)

SECONDARY OUTCOMES:
Screening Time | This will be measured at baseline.
  Use a stopwatch to record the time from the beginning to the end of each measurement tool at baseline . Units of measurement is minutes and seconds
Screening Completion | This will be measured at baseline.
  The screening completion rate is defined as completing the each tool for the frailty screening of the elderly in the community at baseline.
Change in Number of Hospitalization | This will be measured at three months and six months.
  occurence of hospitalization
Change in Number of Falls | This will be measured at three months and six months.
  occurence of falls

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Ru Lin, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Wei Gong Memorial Hospital, Toufen Township, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbasi M, Khera S, Dabravolskaj J, Garrison M, King S. Identification of Frailty in Primary Care: Feasibility and Acceptability of Recommended Case Finding Tools Within a Primary Care Integrated Seniors' Program. Gerontol Geriatr Med. 2019 May 15;5:2333721419848153. doi: 10.1177/2333721419848153. eCollection 2019 Jan-Dec. PMID 31192278
- [Background] Ambagtsheer RC, Thompson MQ, Archibald MM, Casey MG, Schultz TJ. Diagnostic test accuracy of self-reported screening instruments in identifying frailty in community-dwelling older people: A systematic review. Geriatr Gerontol Int. 2020 Jan;20(1):14-24. doi: 10.1111/ggi.13810. Epub 2019 Nov 14. PMID 31729157
- [Background] Fukutomi E, Okumiya K, Wada T, Sakamoto R, Ishimoto Y, Kimura Y, Kasahara Y, Chen WL, Imai H, Fujisawa M, Otuka K, Matsubayashi K. Importance of cognitive assessment as part of the "Kihon Checklist" developed by the Japanese Ministry of Health, Labor and Welfare for prediction of frailty at a 2-year follow up. Geriatr Gerontol Int. 2013 Jul;13(3):654-62. doi: 10.1111/j.1447-0594.2012.00959.x. Epub 2012 Nov 22. PMID 23170783
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Kiely DK, Cupples LA, Lipsitz LA. Validation and comparison of two frailty indexes: The MOBILIZE Boston Study. J Am Geriatr Soc. 2009 Sep;57(9):1532-9. doi: 10.1111/j.1532-5415.2009.02394.x. Epub 2009 Jul 21. PMID 19682112
- [Background] Sutton JL, Gould RL, Daley S, Coulson MC, Ward EV, Butler AM, Nunn SP, Howard RJ. Psychometric properties of multicomponent tools designed to assess frailty in older adults: A systematic review. BMC Geriatr. 2016 Feb 29;16:55. doi: 10.1186/s12877-016-0225-2. PMID 26927924